CLINICAL TRIAL: NCT06339944
Title: Effects of Sensory Motor Training Versus Kinesthetic Exercises on Pain, Range of Motion, Proprioception and Quality of Life in Knee Osteoarthritis .
Brief Title: Effects of Sensory Motor Training and Kinesthetic Exercises in Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR& AHS/23/0198RubabTalib
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; pain; SMT
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sensory motor training along with conventional therapy. (Experimental): This group will receive sensory motor training exercises after the conventional therapy.
  The participants who will be allocated to the SMT group received the same warm-up and stretching program as the CT group, with the same duration and frequency of treatment, but with replacement of the strengthening program with a program emphasizing agility, coordination and balance.
  Interventions: Other: sensory motor training
- kinesthetic exercises along with conventional therapy. (Active Comparator): Group will receive kinesthetic balance exercises after the conventional therapy. All agility-based exercises will be conducted before progressing to balance exercises. For the balance exercises, the participants performed static and dynamic balance exercises with eyes open and then closed by standing on a hard surface and then standing on a soft surface.
  Interventions: Other: kinesthetic exercises

INTERVENTIONS:
Other: sensory motor training — in this group 17 participants will receive conventional therapy and then followed by kinesthetic exercises. 3 sessions per week includes 10 repetitions with 3sets.
  Other Names: conventional therapy
  Arms: sensory motor training along with conventional therapy.
Other: kinesthetic exercises — in this group 17 participants will receive conventional therapy and then followed by kinesthetic exercises. 3 sessions per week includes 10 repetitions with 3sets.
  Other Names: conventional therapy
  Arms: kinesthetic exercises along with conventional therapy.

SUMMARY:
In this study i will see the effects of kinesthetic exercises and sensory motor training on pain and range of motion in patients with knee OA.

DETAILED DESCRIPTION:
In 2022 a A Pilot Randomized Trial of Different Weekly Applications of Kinesthesia, Balance and Agility Exercise Program for Individuals with Knee Osteoarthritis was conducted.In 2023 A critically appraised research was conducted on Sensorimotor or Balance Training to Increase Knee-Extensor and Knee-Flexor Maximal Strength in Patients With Knee Osteoarthritis.

In past there is no study that compares the effects of SMT and kinesthetic exercises in knee OA.

ELIGIBILITY:
Inclusion Criteria:

* patients having osteophytes and definite joint space reduction confirmed by radiographs
* Patients having age 40-60 years or both gender are included

Exclusion Criteria:

Rheumatoid arthritis. Hip or ankle instability Hip or knee replacement Unresolved balance disorder Patients with active synovitis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
VAS | 6th week
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels.

SECONDARY OUTCOMES:
goniometer | 6th week
  a device that measures an angle or permits the rotation of an object to a definite position
WOMAC questionaire | 6th week
  Western Ontario and McMaster Universities (WOMAC) Osteoarthritis index is a multidimensional self-reported disease-specific questionnaire that assesses pain, stiffness and physical disability in patients with Osteoarthritis (OA) of the knee joint. The Swedish version of WOMAC is a reliable, valid, and responsive instrument with metric properties in agreement with the original widely used version.(16
joint position sense test | 6th week
  Joint position sense is one of the most commonly used measures of proprioception.
  Determining JPS involves measuring the accuracy of joint-angle The joint position reproduction test for JPS using goniometry demonstrated moderate to good test-retest reliability and acceptable measurement error in healthy adults.replication,which can be conducted actively or passively and in an open or closed chain environment.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- Tariq Hospital, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] UzunkulaoGlu A, KerIm D, Ay S, ErgIn S. Effects of Single-Task Versus Dual-Task Training on Balance Performance in Elderly Patients With Knee Osteoarthritis. Arch Rheumatol. 2019 Apr 26;35(1):35-40. doi: 10.5606/ArchRheumatol.2020.7174. eCollection 2020 Mar. PMID 32637918
- [Background] Kus G, Tarakci E, Razak Ozdincler A, Ercin E. Sensory-motor training versus resistance training in the treatment of knee osteoarthritis: A randomized controlled trial. Clin Rehabil. 2023 May;37(5):636-650. doi: 10.1177/02692155221137642. Epub 2022 Nov 12. PMID 36373731
- [Background] Gomiero AB, Kayo A, Abraao M, Peccin MS, Grande AJ, Trevisani VF. Sensory-motor training versus resistance training among patients with knee osteoarthritis: randomized single-blind controlled trial. Sao Paulo Med J. 2018 Jan-Feb;136(1):44-50. doi: 10.1590/1516-3180.2017.0174100917. Epub 2017 Dec 7. PMID 29236934